CLINICAL TRIAL: NCT05756322
Title: A Phase 1/2, Open-label, Dose Escalation and Expansion Study to Evaluate the Safety and Tolerability of LBS-007 in Patients With Relapsed or Resistant Acute Leukaemias
Brief Title: The Safety and Tolerability of LBS-007 in Patients With Relapsed or Resistant Acute Leukaemias
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lin BioScience, Inc (Industry)
Collaborators: Lin BioScience Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBS-007-CT01
Record Dates: First submitted 2022-10-20; First posted 2023-03-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Resistant Acute Leukaemias
Keywords: CDC7 inhibitor; LBS-007; AML; ALL
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Finding and Expansion Phase (Experimental): Phase 1: Dose finding phase to evaluate LBS-007 as a monotherapy and combination with Venetoclax and Azacitidine Phase 2: Dose expansion phase to evaluate LBS-007 as a monotherapy and combination therapy at the optimal dose identified by phase 1 (dose finding)
  Interventions: Drug: LBS-007

INTERVENTIONS:
Drug: LBS-007 — Open Label.

SUMMARY:
The most common types of acute leukaemia are acute lymphoblastic leukaemia (ALL) and acute myeloid leukaemia (AML). AML is a heterogenous clonal disorder of haemopoietic progenitor cells and the most common and severe malignant leukemia in adults and is responsible for the highest mortality from leukemia. ALL is a neoplasm characterized by the growth of malignant lymphoblasts of the B or T lineage, leading to an inhibition of proliferation of the normal blood cell lineages.

The primary objectives of this study are investigating the safety, tolerability, and the MTD of LBS-007. The secondary objectives are to assess the efficacy and to determine the pharmacokinetics (PK) of LBS-007. The exploratory objective is to study and correlate the changes in surrogate biomarkers in response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects greater than 18 years old, inclusive.
* Pathologically confirmed diagnoses of Relapsed or resistant AML or ALL.
* Patients who are ineligible for standard therapies that are anticipated to result in durable remission or cure, or who have no known therapy options of documented benefit.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

Exclusion Criteria:

* Concomitant chemotherapy, radiation therapy, or immunotherapy.
* Receiving any other investigational agents concurrently or within 30 days prior to screening.
* Patient has acute promyelocytic leukaemia or leukemia with active CNS involvement.
* History of another active malignancy with 2 years prior to study entry, basal cell skin cancer and previous carcinoma in treated curatively.
* Patient with mental deficits and/or psychiatric history that precludes them from giving informed consent or from following protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number, severity and duration of adverse events (AEs) and treatment-related AEs according to Common Terminology Criteria for Adverse Events (CTCAE) v5. | From baseline through 28 days after end of last treatment cycle (up to 12 months)
Recommended Phase 2 Dose (RP2D) of LBS-007 in the subject population. | From baseline through 28 days after end of last treatment cycle (up to 12 months)

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of LBS-007 in plasma. | Immediately before treatment initiation on Day 1, 3, and 5, or before treatment completion (Day 8), - Then 0.5 (±5 minutes), 1, 2, 4, 6, 10, and 24 (±15 minutes) hours after treatment initiation (Day 1) or completion (Day 8) of first treatment cycle.
Time to Maximum Plasma Concentration (Tmax) of LBS-007 in plasma. | Immediately before treatment initiation on Day 1, 3, and 5, or before treatment completion (Day 8), - Then 0.5 (±5 minutes), 1, 2, 4, 6, 10, and 24 (±15 minutes) hours after treatment initiation (Day 1) or completion (Day 8) of first treatment cycle.
Area under the drug concentration-time curve (AUC) of LBS-007 in plasma. | Immediately before treatment initiation on Day 1, 3, and 5, or before treatment completion (Day 8), - Then 0.5 (±5 minutes), 1, 2, 4, 6, 10, and 24 (±15 minutes) hours after treatment initiation (Day 1) or completion (Day 8) of first treatment cycle.
Efficacy of LBS-007 assessed by bone marrow and peripheral blood. | From baseline through 28 days after end of last treatment cycle (up to 12 months)
  Objective response rate (ORR): Defined for AML as complete response (CR), CR with partial hematological recovery (CRh), CR with incomplete hematological recovery (CRi), morphologic leukemia free state (MLFS), or partial response (PR) as assessed by bone marrow and peripheral blood Defined for ALL as CR, CRh, CRi, or MLFS

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - The University of Kansas Hospital, Fairway, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Australia (6):
  - Wollongong Private Hospital, Wollongong, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - The Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Hollywood Private Hospital, Nedlands, Washington
  - Q Medical Conselling, Perth, Western Australia
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No